CLINICAL TRIAL: NCT00495651
Title: Benefits and Risks of Early Antiretroviral Therapy in HIV-infected Adults in Abidjan, Côte d'Ivoire: Randomized Controlled Trial (ANRS 12136 TEMPRANO)
Brief Title: Early Antiretroviral Treatment and/or Early Isoniazid Prophylaxis Against Tuberculosis in HIV-infected Adults (ANRS 12136 TEMPRANO)
Acronym: TEMPRANO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Gilead Sciences (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 12136 TEMPRANO
Record Dates: First submitted 2007-07-02; First posted 2007-07-03 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: HIV Infections; Tuberculosis
Keywords: HIV; HAART; Early Intervention; Naive patients
MeSH Terms: conditions — HIV Infections; Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- I (Active Comparator): Standard of care
  Interventions: Drug: Antiretroviral medications
- II (Experimental): Standard of care+Isoniazid Prophylaxis:
  Interventions: Drug: Antiretroviral medications+Isoniazid prophylaxis
- III (Experimental): Early Antiretroviral therapy
  Interventions: Drug: Antiretroviral medications
- IV (Experimental): Early Antiretroviral therapy + Isoniazid prophylaxis
  Interventions: Drug: Antiretroviral medications+Isoniazid prophylaxis

INTERVENTIONS:
Drug: Antiretroviral medications — Antiretroviral medications initiation at any time during the trial if at least one WHO-recommended criterion for starting ART is observed.
  Arms: I
Drug: Antiretroviral medications+Isoniazid prophylaxis — * Antiretroviral initiation at any time during the trial if at least one 2009 WHO-recommended criterion for starting ART is observed.
  * Isoniazid prophylaxis:300 mg of INH once a day before breakfast for six months, starting one month after study inclusion
  Arms: II
Drug: Antiretroviral medications — Early ART initiation on the day of inclusion, before reaching the current WHO criteria
  Arms: III
Drug: Antiretroviral medications+Isoniazid prophylaxis — * Early Antiretroviral medications initiation on the day of inclusion, before reaching the current WHO criteria
  * Isoniazid prophylaxis: 300 mg of INH once a day before breakfast for six months, starting one month after study inclusion
  Arms: IV

SUMMARY:
The Temprano trial is based on the following assumptions:

* ART initiation at CD4 counts <800/mm3 could significantly reduce the probability of severe HIV-related morbidity or death in the medium term.
* Tuberculosis and tuberculosis-related deaths are likely to represent a considerable proportion of morbidity and mortality among HIV-infected patients with high CD4 counts in sub-Saharan Africa. Therefore, 6-month Isoniazide Prophylaxis for Tuberculosis (IPT) and early ART could enhance each others efficacy.

DETAILED DESCRIPTION:
* The main individual benefit of very early ART initiation is likely a reduction in early severe AIDS-defining and non-AIDS-defining morbidity. While the diseases that might justify earlier initiation in high-income countries are generally non-infectious (non-AIDS-defining malignancies, renal diseases and cardiovascular diseases), the leading cause of early severe AIDS-defining morbidity in sub-Saharan Africa is tuberculosis and the main causes of severe non-AIDS-defining morbidity are non-invasive bacterial diseases. As a result of poor access to diagnosis and care, some HIV-infected people die from early infectious diseases before reaching current WHO criteria for starting ART.
* Although the Côte d'Ivoire National Tuberculosis Program (PNLT) does not authorize the use of prophylaxis against tuberculosis, it has allowed the Temprano trial to provide a six-month course of isoniazid (INH) prophylaxis to half of the study subjects. This will allow us to (i) put early ART in perspective with a early 6-month INH prophylaxis use, in a setting where tuberculosis is the first cause of severe HIV-associated morbidity; and (ii) to describe and assess the feasibility of a six-month course of INH prophylaxis among patients with high CD4 counts.
* Some drug toxicities are immediate but reversible. If early ART is compared to no ART in the short term, these toxicities may demonstrate erroneously that early ART is unfavorable. The risks and benefits of early ART initiation should therefore be evaluated over the long term. In the Temprano trial, we will: (i) follow patients for at least 30 months and analyze the primary outcome at 30 months; (ii) follow some study subjects for 80 months and evaluate the evolution of the ART efficacy / toxicity ratio from month 30 to month 80 as a secondary endpoint, to inform future policies if early ART is found to be beneficial at 30 months.

Main objective: To assess the benefits and risks of starting ART immediately and/or to receive a 6-month IPT among HIV-infected adults with CD4 counts <800mm3 and no criteria for starting ART immediately according to the most recent WHO guidelines.

Location: Abidjan, Côte d'Ivoire.

Methods: randomized 2x2 factorial superiority trial

Main inclusion criteria: (i) HIV-1 or HIV-1+2 infection; (ii) age >18 years; (iii) nadir CD4 count <800/mm3 and no criteria for starting ART immediately according to the most recent WHO guidelines; and (iv) no active tuberculosis.

Trial arms: Arm I: ART initiation according to WHO criteria, at any time during follow-up; Arm II: INH prophylaxis (300 mg/day) for six months and ART initiation according to WHO criteria, at any time during follow-up; Arm III: immediate ART initiation, before reaching the WHO criteria; Arm IV: INH prophylaxis (300 mg/day) for six months and immediate ART initiation, before reaching the WHO criteria.

First-line ART regimens

* Tenofovir / emtricitabine + efavirenz for all HIV-1-infected men and all HIV-1-infected women who meet the following requirements: on effective contraception and no history of nevirapine use for the prevention of mother-to-child transmission of HIV (PMTCT).
* Tenofovir / emtricitabine + lopinavir / ritonavir for all HIV-1+2-infected patients and all women who do not use effective contraception or who have a history of nevirapine use for PMTCT.

Primary endpoint: Death (all-cause), AIDS-defining disease, non-AIDS-defining malignancy, or non-AIDS-defining invasive bacterial disease.

Main secondary endpoint: Grade 3 or 4 clinical event (including renal and cardiovascular events) or laboratory test result, as defined by the ANRS classification system of drug-related adverse events.

Final primary analysis: It will be performed once the last patient has reached 30 months of follow-up. Time-dependent analyses will compare the primary outcome : (i) among patients initiating ART immediately (arms III and IV) versus patients initiating ART according to the WHO criteria (arms I and II); (ii) among patients who were prescribed a 6-months (arms II and IV) IPT versus those who were not (arms I and III).

Intermediate analysis on safety criteria:

* Toxicity: all-cause mortality. We have not planned to perform any intermediate analyses for this criterion. If the number of observed deaths is higher than anticipated, however, the DSMB may decide to carry one out. In this case, we will adjust the alpha coefficient using the method suggested by Pocock to account for the large variety of available tests.
* Efficacy: incidence of severe morbidity. Intermediate analysis: We have not planned any intermediate analyses for this criterion. If the number of severe morbidity evens is higher than anticipated once all patients have reached 12 months of follow-up, the DSMB may decide to carry one out. In this case, we will adjust the alpha coefficient using the method suggested by Haybittle-Peto, to account for the large variety of available tests.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 or HIV-1 + HIV-2 infection
* Age >18 years
* No ongoing active tuberculosis
* Home address in any district of the greater Abidjan area
* Written informed consent before any clinic visit or laboratory test
* Clinical and immunologic status:CD4 counts <800/mm3 and no criteria for starting ART according to the most recent WHO guidelines

Exclusion Criteria:

* Pregnant or breastfeeding women
* HIV-2 infection alone
* Clinical signs suggesting a severe disease (including tuberculosis) that has not yet been diagnosed, such as fever, wasting, diarrhea or unexplained cough (partial list)
* Previous ART initiation
* Known severe renal, cardiac or hepatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2073 (Actual)
Dates: Start 2008-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Death (all-cause), or severe HIV-related disease (AIDS-defining diseases, non-AIDS-defining malignancies, and non-AIDS-defining invasive bacterial diseases) | 30 months
  * Severe HIV-related disease are defined as AIDS-defining diseases, non-AIDS- defining malignancies, and non-AIDS-defining invasive bacterial diseases
  * Invasive bacterial diseases are defined as: bacteremia, or bacterial infection of any solid organ or aseptic cavity (eg: pneumonia, pleurisy, meningitis,pyomyositis, pyelonephritis, prostatitis, orchitis, epididymitis, salpingitis, endometritis, endocarditis, cholecystitis, visceral abscesses).
prevalence of HIV resistance (ANRS12253 associated study) | 30 month after ARV initiation

SECONDARY OUTCOMES:
Grade 3 or 4 clinical events (including cardiovascular, renal and bone disease) and laboratory test results, as defined by the ANRS classification system of drug-related adverse events | 30 months
Tuberculosis disease or tuberculosis-related death | 30 months
Changes in CD4 counts | 30 months
Resistance to antiretroviral medications | 30 months
Adherence to treatment | 30 months
Individual socio-economic factors | 30 months
Quality of life | 30 months
Conversions and reversions of repeated QuantiFERON® TB Gold tests between inclusion and month 12 (M12)(ANRS12224 associated study) | 12 months
Cost-effectiveness of each trial arm in the short- and long-term | 30 months
Death | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Anglaret, MD, PhD, Principal Investigator — Université Bordeaux 2; Serge Eholié, MD, MSc, Pr, Principal Investigator — CHU de Treichville, Abidjan
Locations (9):
- Côte d’Ivoire (9):
  - Centre de prise en charge de personnes vivant avec le VIH la pierre angulaire, Abidjan
  - Centre de Prise en Charge et de Formation ACONDA, Abidjan
  - Centre de Suivi des donneurs de sang, Centre National de Transfusion Sanguine, Abidjan
  - Centre Intégré de Recherches Biocliniques d'Abidjan, Abidjan
  - Centre médico-social El Rapha, Abidjan
  - Formation Sanitaire Urbaine Anonkoua Kouté, Abidjan
  - Hopital Général Felix Houphouet Boigny, Abidjan
  - Service des Maladies Infectieuses et Tropicales, CHU de Treichville, Abidjan
  - Unité de Soins Ambulatoires et de Conseil, CHU de Treichville, Abidjan

REFERENCES:
- [Derived] Moh DR, Ntakpe JB, Gabillard D, Yayo-Emieme AA, Badje A, Kouame GM, d'Aquin TT, Danel C, Anglaret X, Eholie SP. Association of cellular HIV-1 DNA and virological success of antiretroviral treatment in HIV-infected sub-Saharan African adults. BMC Infect Dis. 2022 Jan 29;22(1):100. doi: 10.1186/s12879-022-07082-2. PMID 35093007
- [Derived] Moh R, Badje A, N'takpe JB, Kouame GM, Gabillard D, Ouassa T, Ouattara E, Le Carrou J, Bohoussou F, Messou E, Eholie S, Anglaret X, Danel C. Screening for active tuberculosis before isoniazid preventive therapy among HIV-infected West African adults. Int J Tuberc Lung Dis. 2017 Dec 1;21(12):1237-1244. doi: 10.5588/ijtld.17.0016. PMID 29297443
- [Derived] Kouame GM, Boyd A, Moh R, Badje A, Gabillard D, Ouattara E, Ntakpe JB, Emieme A, Maylin S, Chekaraou MA, Eholie SP, Zoulim F, Lacombe K, Anglaret X, Danel C; French National Agency for Research on AIDS and Viral Hepatitis (ANRS) 12136 Temprano and ANRS 12240 VarBVA Study Groups. Higher Mortality Despite Early Antiretroviral Therapy in Human Immunodeficiency Virus and Hepatitis B Virus (HBV)-Coinfected Patients With High HBV Replication. Clin Infect Dis. 2018 Jan 6;66(1):112-120. doi: 10.1093/cid/cix747. PMID 29020361
- [Derived] TEMPRANO ANRS 12136 Study Group; Danel C, Moh R, Gabillard D, Badje A, Le Carrou J, Ouassa T, Ouattara E, Anzian A, Ntakpe JB, Minga A, Kouame GM, Bouhoussou F, Emieme A, Kouame A, Inwoley A, Toni TD, Ahiboh H, Kabran M, Rabe C, Sidibe B, Nzunetu G, Konan R, Gnokoro J, Gouesse P, Messou E, Dohoun L, Kamagate S, Yao A, Amon S, Kouame AB, Koua A, Kouame E, Ndri Y, Ba-Gomis O, Daligou M, Ackoundze S, Hawerlander D, Ani A, Dembele F, Kone F, Guehi C, Kanga C, Koule S, Seri J, Oyebi M, Mbakop N, Makaila O, Babatunde C, Babatounde N, Bleoue G, Tchoutedjem M, Kouadio AC, Sena G, Yededji SY, Assi R, Bakayoko A, Mahassadi A, Attia A, Oussou A, Mobio M, Bamba D, Koman M, Horo A, Deschamps N, Chenal H, Sassan-Morokro M, Konate S, Aka K, Aoussi E, Journot V, Nchot C, Karcher S, Chaix ML, Rouzioux C, Sow PS, Perronne C, Girard PM, Menan H, Bissagnene E, Kadio A, Ettiegne-Traore V, Moh-Semde C, Kouame A, Massumbuko JM, Chene G, Dosso M, Domoua SK, N'Dri-Yoman T, Salamon R, Eholie SP, Anglaret X. A Trial of Early Antiretrovirals and Isoniazid Preventive Therapy in Africa. N Engl J Med. 2015 Aug 27;373(9):808-22. doi: 10.1056/NEJMoa1507198. Epub 2015 Jul 20. PMID 26193126
- [Derived] Danel C, Kabran M, Inwoley A, Badje A, Herrmann JL, Moh R, Lecarrou J, Gabillard D, Ntakpe JB, Deschamps N, Ouattara E, Perronne C, Eholie S, Anglaret X. Quantiferon-TB Gold: performance for ruling out active tuberculosis in HIV-infected adults with high CD4 count in Cote d'Ivoire, West Africa. PLoS One. 2014 Oct 16;9(10):e107245. doi: 10.1371/journal.pone.0107245. eCollection 2014. PMID 25330161
- [Derived] Jean K, Gabillard D, Moh R, Danel C, Desgrees-du-Lou A, N'takpe JB, Le Carrou J, Badje A, Eholie S, Lert F, Anglaret X, Dray-Spira R. Decrease in sexual risk behaviours after early initiation of antiretroviral therapy: a 24-month prospective study in Cote d'Ivoire. J Int AIDS Soc. 2014 Jun 30;17(1):18977. doi: 10.7448/IAS.17.1.18977. eCollection 2014. PMID 24985779
- [Derived] Ouattara E, Danel C, Moh R, Gabillard D, Peytavin G, Konan R, Carrou JL, Bohoussou F, Eholie SP, Anglaret X. Early upper digestive tract side effects of zidovudine with tenofovir plus emtricitabine in West African adults with high CD4 counts. J Int AIDS Soc. 2013 Apr 30;16(1):18059. doi: 10.7448/IAS.16.1.18059. PMID 23639243
- See also: Related Info — http://www.anrs.fr
- See also: ANRS 12136 Temprano trial website — http://mereva.net/temprano